CLINICAL TRIAL: NCT03510832
Title: Evaluation of Antithrombotic STrategies in STEMI Patients in China
Acronym: EAST-STEMI
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Qilu Hospital of Shandong University (Other)
Collaborators: Shandong Provincial Hospital (Other Government); Qianfoshan Hospital (Other); Jinan Central Hospital (Other); The Second Hospital of Shandong University (Other); Shandong Province Third hospital (Other); The 5th People's Hospital of Jinan (Unknown); The 6th People's Hospital of Jinan (Unknown); The Affiliated Hospital of Qingdao University (Other); Qingdao Municipal Hospital (Other); Qingdao Central Hospital (Other); Qingdao Haici Hospital (Other); Chengyang People's Hospital (Unknown); Qingdao Westcoast New Area Central Hospital (Unknown); Qingdao Jiaozhou Central Hospital (Unknown); Pingdu People's Hospital (Unknown); Central Hospital of Zibo (Other); Zibo First Hospital (Other); Linzi District People's Hospital (Unknown); Peking University Care Luzhong Hospital (Other); Tengzhou Central People's Hospital (Other Government); Dongying People's Hospital (Other); Shengli Oilfield Hospital (Other); Yantaishan Hospital (Unknown); Yantai Yuhuangding Hospital (Other); Yantai Affiliated Hospital of Binzhou Medical University (Other); Longkou People's Hospital (Unknown); Laizhou City People's Hospital (Other); Weifang People's Hospital (Other); Weifang Medical University (Other); Weifang Traditional Chinese Hospital (Unknown); Yidu Central Hospital of Weifang (Unknown); Qingzhou People's Hospital (Unknown); Shouguang people's Hospital (Unknown); Jining Medical University (Other); Jining First People's Hospital (Other); Wenshang People's Hospital (Unknown); Yanzhou Branch of Affiliated Hospital of Jining Medical University (Unknown); Jinxiang People's Hospital (Unknown); Taian City Central Hospital (Other); Taishan Medical University Affiliated Hospital (Other); Feicheng People's Hospital (Unknown); Weihai Municipal Hospital (Other); Weihai Central Hospital (Other); Binzhou Medical University (Other); Zhouping People's Hospital (Unknown); Dezhou People's Hospital (Other); Ningjin County People's Hospital (Unknown); Liaocheng People's Hospital (Other); The Second People's Hospital of Liaocheng (Unknown); Linyi People's Hospital (Other); Feixian People's Hospital (Unknown); Heze Municipal Hospital (Other); Yuncheng County People's Hospital (Unknown); Heze Luxin Cardiovascular and Cerebrovascular Hospital (Unknown); Jining Integrative Medicine Hospital (Unknown); Tianjin Chest Hospital (Other); Henan Provincial People's Hospital (Other); Inner Mongolia People's Hospital (Other); Anhui Provincial Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: QLEmer201802
Record Dates: First submitted 2018-03-20; First posted 2018-04-27 (Actual); Last update posted 2018-04-27 (Actual); Status verified 2018-03

CONDITIONS: STEMI; Emergent PCI
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- STEMI patients undergoing Emergent PCI

SUMMARY:
EAST-STEMI is the first perspective, multicenter, large-scale registry focusing on the evaluation of real-world medical quality (especially PCI quality) and antithrombotic strategies in STEMI patients undergoing emergent PCI in a regional representative sample in China with 2 years follow-up. Clinical decision support tools (including ischemic score, bleeding score, etc) will be developed and validated based on the database. Novel biomarkers to predict the prognosis and to support risk stratification will be explored by using the blood samples.

ELIGIBILITY:
Inclusion Criteria:

1. Age>=18yrs
2. STEMI patients undergoing emergent PCI
3. Signed informed consent

Exclusion Criteria:

1. Difficult to follow up or obtain accurate information (e.g., long-term overseas stay, speech or mental disorders)
2. Other severe diseases (e.g., liver failure, renal failure and advanced stage of cancer)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: consecutive STEMI patients undergoing emergent PCI
Sampling Method: Non-Probability Sample
Enrollment: 8000 (Estimated)
Dates: Start 2018-03-01 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Net Adverse Clinical Events (NACEs) | 2 years after emergent PCI
  The primary outcome is the rate of adjudicated NACEs, a composite of major adverse cardiac or cerebral events (MACCEs) and bleeding. MACCEs include cardiac death, reinfarction, urgent revascularization, or stroke. Bleeding is defined by the Bleeding Academic Research Consortium (BARC) definition (types 1-5). BARC type 2 bleeding is considered as minor bleeding, type 3-5 bleeding is considered as major bleeding.

SECONDARY OUTCOMES:
Contrast-induced acute kidney injury (CI-AKI) | 72 hours after contrast exposure
  CI-AKI is defined as an increase in serum creatinine of ≥0.3mg/dl or ≥50% from baseline within 72 hours.
Definite/Probable Stent thrombosis | 2 years after emergent PCI
  Stent thrombosis is defined according to the Academic Research Consortium criteria. Definite stent thrombosis is defined as angiography or autopsy examination confirmed stent occlusion or thrombus. Probable stent thrombosis is defined as death occurring within 30 days that cannot be attributed to another cause or when myocardial infarction occurs at any time point and is attributable to the target vessel in the absence of angiography confirming another culprit lesion.
Heart failure | 2 years after emergent PCI
  Heart failure is defined as physician documentation or report of any of the following clinical symptoms of heart failure described as unusual dyspnea on light exertion, recurrent dyspnea occurring in the supine position, fluid retention; or the description of rales, jugular venous distension, pulmonary edema on physical exam, or pulmonary edema on chest x-ray. A low ejection fraction alone, without clinical evidence of heart failure does not qualify as heart failure.
Quality of life (QoL) | 2 years after emergent PCI
  QoL is assessed by using EuroQol-5 Dimension (EQ-5D), which is the most widely used generic instrument to measure QoL. The utility index scores of EQ-5D represent the QoL.The higher the score, the better the QoL.

CONTACTS AND LOCATIONS:
Overall Officials: Yuguo Chen, Dr, Principal Investigator — Qilu Hospital of Shandong University
Locations (1):
- Qilu Hospital of Shandong University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No